CLINICAL TRIAL: NCT00787722
Title: Trial of High Dose Immunosuppressive Therapy With Hematopoietic Stem Cell Support in Devic's Disease
Brief Title: Hematopoietic Stem Cell Transplant in Devic's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD Devic's Disease Auto 2008
Record Dates: First submitted 2008-10-31; First posted 2008-11-07 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-11

CONDITIONS: Devic's Disease
Keywords: High dose immunosuppressive therapy; Hematopoietic stem cell support
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Hematopoietic Stem Cell Transplantation; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; thymoglobulin; Antilymphocyte Serum; Mesna; Rituximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Hematopoietic stem cell transplantation will be performed after conditioning regimen of cyclophosphamide, G-CSF, Mesna, rATG, rituximab, and methylprednisolone.
  Interventions: Procedure: Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: G-CSF; Drug: rATG; Drug: Mesna; Drug: Rituximab; Drug: Methylprednisolone

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplantation — Infusion of participant's own stem cells
Drug: Cyclophosphamide — A medication used as chemotherapy and to suppress the immune system
  Other Names: Cytoxan; Neosar
Drug: G-CSF — A glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Drug: rATG — A rabbit polyclonal antibody to lymphocytes
  Other Names: Thymoglobulin; Anti-Thymocyte Globulin
Drug: Mesna — A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  Other Names: Mesnex
Drug: Rituximab — Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Other Names: Rituxan
Drug: Methylprednisolone — A corticosteroid medication used to suppress the immune system and decrease inflammation
  Other Names: Solu-Medrol; Depo-Medrol

SUMMARY:
This study is designed to examine whether treating Devic's disease patients with high dose cyclophosphamide together with rabbit antithymocyte globulin (rATG)/rituximab (drugs which reduce the function of the immune system), followed by return of previously collected patient's stem cells will result in improvement in Devic's disease. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the intense chemotherapy is to destroy the cells in patient's immune system, which may be causing his/her disease. The purpose of the stem cell infusion is to produce a normal immune system that will no longer attack patient's body. The purpose of study is to examine the safety and efficacy of this treatment. The drugs used in this study treatment are drugs for commonly used for immune suppression.

DETAILED DESCRIPTION:
Neuromyelitis optica (NMO, Devic's disease) is an autoimmune, inflammatory, demyelinating central nervous system disorder in which a person's own immune system attacks the optic nerves and spinal cord and is characterized by concurrence of optic neuritis and transverse myelitis, typically associated with a lesion in the spinal cord extending over three or more vertebral segments. Although it is most commonly relapsing, it is distinct from multiple sclerosis in that it is more severe, tends to spare the brain, and is associated with a longitudinally extensive lesion on spinal cord MRI. Furthermore, NMO is associated with a highly specific serum autoantibody marker, NMO-immunoglobulin G (IgG), which targets the water channel aquaporin-4. The disease follows a relapsing course in more than 90% of patients.

At present, parenteral corticosteroids are widely employed as first-line treatment of optic neuritis and myelitis attacks, whereas therapeutic plasmapheresis is applied in the case of corticosteroids failure. Various strategies for the prevention of NMO relapses have been employed in small case series with modest activity. Immune based therapies, in order to be effective, need to be started early in the disease course while Devic's disease is predominantly an immune-mediated and inflammatory disease. Since 50% of patients with NMO are confined to a wheelchair within 5 years of onset, new therapies are needed in this disease.

We now propose, as a phase I study, complete immune ablation and subsequent reconstitution with autologous stem cells.

Based on the experience of the pilot studies, the current protocol will mobilize stem cells with granulocyte-colony stimulating factor (G-CSF) and cyclophosphamide and collect stem cells by apheresis. A subsequent bone marrow harvest will be performed only if needed to supplement the peripheral blood stem cells (PBSC). Based on experience of autoimmune flares in patients receiving G-CSF alone for mobilization, patients will be mobilized with cyclophosphamide 2.0 g/m2 and G-CSF 5- 10 mcg /kg.

In order to avoid cumulative cardiac toxicity from cyclophosphamide and to allow culture of hematopoietic stem cell (HSC) product, three weeks must separate the administration of cyclophosphamide for mobilization and for conditioning.

Cyclophosphamide 50 mg/kg/day will be given IV over 2 hours in 500 cc of normal saline. If actual weight is < ideal weight, cyclophosphamide will be given based on actual weight. If actual weight is > ideal weight, cyclophosphamide will given as adjusted weight. Adjusted weight = ideal weight + 25% (actual weight minus ideal weight).

Hydration-guidelines, normal saline (NS) at 150-200 ml/hr should be given 2 hours before cyclophosphamide and continued until 24 hours after the last cyclophosphamide dose. The rate of hydration will be aggressively adjusted. Twice daily weights will be obtained. Amount of fluid can be modified based on patient's fluid status.

r ATG 0.5 mg/kg given on day -5, then 1.0 mg/kg given on day -4, then 1.5 mg/kg given on days -3 through -1. rATG is infused over 10 hours. Premedicate with Acetaminophen 650 mg po and Diphenhydramine 25 mg po/IV 30 minutes before the infusion.

Rituxan ( Rituximab ) - The dose of 500 mg of Rituximab will be diluted in 500 ml 0.9 % NS and infused per standard Rituximab infusion guidelines, given on days -6 and on day + 1. Following the guidelines, Rituximab will be started at 50 mg/hr. If no reaction occurs, the dose will be increased by 50 mg/hr every 30 minutes to a maximum of 400 mg/hr.

G-CSF - guidelines, 5-10 mcg/kg/day will be started day + 5 and continued until the absolute neutrophil counts reaches at least 1,000/µl.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16-65, at the time of pretransplant evaluation
* An established diagnosis of Devic's disease (more than one acute attack)
* NMO- IgG aquaporin-4 autoantibody positive

Exclusion Criteria:

* Paraplegia or quadriplegia and legal blindness (defined as visual acuity of 20/200 or less in the better eye with the best correction possible)
* Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy
* Prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix. Other malignancies for which the patient is judged to be cured, such as head and neck cancer, or breast cancer will be considered on an individual basis
* Positive pregnancy test
* Inability or unwillingness to pursue effective means of birth control. Effective birth control is defined as 1) refraining from all acts of vaginal intercourse (ABSTINENCE); 2) consistent use of birth control pills; 3) injectable birth control methods (Depo-provera, Norplant); 4) tubal sterilization or male partner who has undergone vasectomy; 5) placement of an intrauterine device (IUD); or 6) use, with every act of intercourse, of diaphragm with contraceptive jelly and/or condoms with contraceptive foam
* Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
* forced expiratory volume at one (FEV1) / forced vital capacity (FVC) < 60% of predicted after bronchodilator therapy (if necessary)
* Diffusing capacity of lung for carbon monoxide (DLCO) < 50% of predicted
* Resting left ventricular ejection fraction (LVEF) < 50 %
* Serum creatinine > 2.0 mg/dl
* Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins
* Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams
* Bilirubin > 2.0 mg/dl
* Platelet count < 100,000/ul or absolute neutrophil count (ANC) < 1000/ul
* Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible
* Active infection except asymptomatic bacteriuria
* Inability to give informed consent
* HIV positive
* Transaminases > 3x of normal limits, liver cirrhosis

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burt RK, Balabanov R, Han X, Burns C, Gastala J, Jovanovic B, Helenowski I, Jitprapaikulsan J, Fryer JP, Pittock SJ. Autologous nonmyeloablative hematopoietic stem cell transplantation for neuromyelitis optica. Neurology. 2019 Oct 29;93(18):e1732-e1741. doi: 10.1212/WNL.0000000000008394. Epub 2019 Oct 2. PMID 31578302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: survival rate will be evaluated at 6 months,1 year, 2 year, 3 year, 4 year, 5 year after the transplant
Time Frame: 6 months, 1 year, 2 year, 3 year, 4 year, 5 year - after the transplant
Population: The reason that the number analyzed in one or more rows differs from the overall number analyzed is because one patient with coexistent SLE died of complications from active lupus 10 months after the transplant and another patient was only 3 years out from transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 13
Participants
  6 months survival | 13
  1 year survival: number analyzed (Participants) | 12
  1 year survival | 12
  2 year survival: number analyzed (Participants) | 12
  2 year survival | 12
  3 year survival: number analyzed (Participants) | 11
  3 year survival | 11
  4 year survival: number analyzed (Participants) | 11
  4 year survival | 11
  5 year survival: number analyzed (Participants) | 11
  5 year survival | 11

2. Secondary Outcome: Quality of Life (QOL) Short Form - 36 (SF-36)
Description: SF- 36 is a self-administered quality of life exam. The evaluation of the results was done by attributing scores to each question, which were then transformed into a scale ranging from 0 to 100, where 0 corresponds to the worst quality of life and 100 to the best.
Time Frame: pre-transplant 12mo and 5 years
Population: The reason that the number analyzed differs in one or more rows is because 1 patient did not complete the form and was excluded. Another patient was not 5 years out from transplant so there is no 5 year data on the patient.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 11
score on a scale
  Pretransplant | 30.83 (34.22)
  1 Year Post Transplant | 52.69 (55.08)
  5 Year Post Transplant: number analyzed (Participants) | 10
  5 Year Post Transplant | 61.63 (62.09)

3. Secondary Outcome: Post HSCT Immune -Modulating Medication and Relapse
Description: Number of immune - modulating medication and relapse evaluated 5 year - after the transplant
Time Frame: Pre transplant and 6 months, 1 year, 2 year, 3 year, 4 year and 5 year after transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Hematopoietic Stem Cell Transplantation (HSCT): Hematopoietic stem cell transplantation will be performed after conditioning regimen of cyclophosphamide, G-CSF, Mesna, rATG, rituximab, and methylprednisolone.
  Hematopoietic Stem Cell Transplantation: Infusion of participant's own stem cells
  Cyclophosphamide: A medication used as chemotherapy and to suppress the immune system
  G-CSF: A glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  rATG: A rabbit polyclonal antibody to lymphocytes
  Mesna: A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  Rituximab: Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Methylprednisolone: A corticosteroid medication used to suppress the immune system and decrease inflammation
Arm/Group | Hematopoietic Stem Cell Transplantation (HSCT)
Number analyzed (Participants) | 12
Participants
  Pre HSCT - Immunosuppression/Relapse Rate | 12
  6 Mos Post HSCT Immunosuppression/ Relapse Rate | 1
  1 Year Post HSCT Immunosuppression/Relapse Rate: number analyzed (Participants) | 11
  1 Year Post HSCT Immunosuppression/Relapse Rate | 1
  2 Year Post HSCT Immunosuppression/Relapse Rate | 3
  3 Year Post HSCT Immunosuppression/Relapse Rate: number analyzed (Participants) | 11
  3 Year Post HSCT Immunosuppression/Relapse Rate | 0
  4 Year Post HSCT Immunosuppression/Relapse Rate: number analyzed (Participants) | 11
  4 Year Post HSCT Immunosuppression/Relapse Rate | 1
  5 Year Post HSCT Immunosuppression Relapse Rate: number analyzed (Participants) | 11
  5 Year Post HSCT Immunosuppression Relapse Rate | 1

4. Secondary Outcome: Number of Patients Who Require No Device Assistance for Ambulation
Description: No Device Assistance Needed for Ambulation evaluated at 6 months, 1 year, 2 year, 3 year, 4 year, 5 year - after the transplant
Time Frame: 6 months, 1 year, 2 year, 3 year, 4 year, 5 year - after the transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 12
Participants
  Pre HSCT- No Assistive Required | 6
  6 Mos Post HSCT- No Assistive Device Required | 9
  1 Year Post HSCT- No Assistive Device Required | 10
  2 Year Post HSCT- No Assistive Device Required | 9
  3 Year Post HSCT- No Assistive Device Required: number analyzed (Participants) | 11
  3 Year Post HSCT- No Assistive Device Required | 8
  4 Year Post HSCT- No Assistive Device Required | 8
  5 Year Post HSCT- No Assistive Device Required: number analyzed (Participants) | 11
  5 Year Post HSCT- No Assistive Device Required | 9

5. Secondary Outcome: Disability Score: Expanded Disability Status Scale (EDSS)
Description: Disability scores (disease improvement defined by at least a 1 point increase in the Expanded Disability Status Scale (EDSS) on consecutive evaluations at least three months apart.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Time Frame: pretransplant 6 month, 5 year
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 13
score on a scale
  Pretransplant Disability Score (EDSS) | 4.4 [2.0 to 6.5]
  1 Year Post Transplant Disability Score (EDSS): number analyzed (Participants) | 12
  1 Year Post Transplant Disability Score (EDSS) | 2.8 [1 to 6.5]
  5 Year Post Transplant Disability Score (EDSS): number analyzed (Participants) | 11
  5 Year Post Transplant Disability Score (EDSS) | 3.3 [0 to 6.5]

6. Secondary Outcome: NMO-IgG Aquaporin- 4 Autoantibody Titer
Description: NMO-IgG aquaporin- 4 autoantibody titer will be tested pretransplant and post transplant.
Time Frame: Pretransplant and 5 year Post Transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 13
Participants
  Pretransplant NMO ASSAY positive: number analyzed (Participants) | 12
  Pretransplant NMO ASSAY positive | 11
  5 year post transplant NMO Assay positive: number analyzed (Participants) | 11
  5 year post transplant NMO Assay positive | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=13)
Unrelated Complications from Systemic Lupus Erythematosus (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=13)
Infection (Infections and infestations) | 1 (1) — C.Diff
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (9) — hypophosphatemia
Neutropenic Fevers (General disorders) | 5 (5) — Neutropenic Fevers
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) — hypocalcemia
Nausea and Vomiting (Metabolism and nutrition disorders) | 3 (3) — nausea and vomiting
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) — hypokalemia
Orthostatic Hypotension (General disorders) | 2 (2) — orthostatic hypotension
Hypertension, Hyperglycemia, Diarrhea (General disorders) | 1 (1) — hypertension, hyperglycemia and diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT00787722/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT00787722/SAP_001.pdf